CLINICAL TRIAL: NCT04656093
Title: Self-management Behaviors Among COPD Patients With Multi-Morbidity
Brief Title: Healthy Mediation Adherence To Transform and Effectively Relieve Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Northwestern University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Juan P Wisnivesky, Chief Of Division of General Internal Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 14-0666; 5R01HL126508-05 (NIH)
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: COPD; Diabetes; Hypertension
Keywords: COPD; Intervention; Motivational Interviewing; Cognitive Restructuring; Diabetes; Hypertension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Intervention Model Description: The study team will use data from the observational component of the study to identify patients with COPD, Diabetes (DM) and/or Hypertension (HTN).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research coordinators (RCs) and Principal Investigator (Juan Wisnivesky) are blinded to study randomization and treatment arm for each participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group - Cognitive Restructuring, Motivational Interviewing, and Multi-Medication Adherence.
  The pilot intervention is comprised of three educational sessions for individual study patients, conducted by interventionist with a master's degree in psychology with cognitive behavioral therapy training. The topics addressed in the sessions are as follows:
  Review of COPD medication inhaler technique, psychoeducation on maladaptive beliefs and emotional response.
  Interventions: Behavioral: Education on SMB; Behavioral: Psychoeducation on ATs for maladaptive beliefs (if applicable); Behavioral: Psychoeducation on emotional response (if applicable)
- Control (Active Comparator): Control group - Supportive counseling for comorbidity management
  Interventions: Behavioral: Supportive counseling

INTERVENTIONS:
Behavioral: Supportive counseling — Participants in the control arm will receive 3 "placebo" sessions to control for the potentially confounding effect of personalized attention from the care coach on the relationship between the intervention and outcomes. The interventionist will review a patient education booklet for COPD self-management over the 3 sessions and address any question raised by the study subject.
  Arms: Control
Behavioral: Education on SMB — Goal is to educate patient on SMB based on responses during 15-month interview and screener call, and assess patient's motivation for change.
  Arms: Intervention
Behavioral: Psychoeducation on ATs for maladaptive beliefs (if applicable) — Goal is to educate patient on relationship between thoughts and SMB, and identify maladaptive beliefs, automatic thoughts, and cognitive distortions.
  Arms: Intervention
Behavioral: Psychoeducation on emotional response (if applicable) — Goal is to educate patient on relationship between emotions and COPD + SMB, identify
  Arms: Intervention

SUMMARY:
The goal of the parent R01 study has been to determine how beliefs about chronic illness and their treatments affect SMB in the context of chronic obstructive pulmonary disease (COPD) with comorbid hypertension (HTN) and or diabetes (DM). The educational counseling modules the study team plans to pilot test are rooted in the Self-Regulation Model (SRM), a theory of health behaviors that has been used to develop interventions, but has only been applied to research on behaviors around single diseases.

DETAILED DESCRIPTION:
Outcomes for patients with multimorbidity (MM) are often poor, in part because of low adherence to self-management behaviors (SMB). Research has identified key determinants of SMB for individual diseases and shown the powerful influence that illness representations and medication beliefs have on these behaviors. Yet, little is known about the impact of illness representations in the context of MM where beliefs about one illness and its treatments may be at odds, or symbiotic, with those for comorbidities. Without this knowledge, ability to provide optimal self-management support for MM patients is limited. The Pilot will be focusing on three mayor components with the hopes to provide optimal self-management support for MM patients:

i. Beliefs about Multi-Morbidity The Care Coach will discuss the participant's individual disease & self-management-related beliefs. This discussion will be guided by a semi-structured questionnaire covering domains from Brief Illness Perception Questionnaire (BIPQ) and the Beliefs about Medication Questionnaire (BMQ) for each pertinent multi-morbidity.

For example, the Care Coach will ask: "How long do you believe that your COPD will continue?" "And how about your hypertension, how long will it continue?" The Care Coach will note the participants' responses to each question, and mark which beliefs seem to be potentially counterproductive to self-management (e.g. very concerned about taking DM medications long-term). These beliefs will be used to focus the intervention session section on cognitive restructuring. Beliefs will be addressed using a Cognitive restructuring approach.

ii. Emotional Response Next, the Care Coach will ask the participant about the role of emotional responses and mental state in their disease management. This will consist of 1-2 semi-structured questions about symptoms of anxiety and depression, as well as the emotional impact of each comorbidity in the participant's life.

For example: "Does your COPD affect you emotionally? [If yes] In what ways?" The Care Coach will take notes on the participants' self-reported emotional response to their comorbidities, as well as any observed indications of distress/emotional reaction to their illnesses. This information, combined with the participants' data from the 15-month DISH interview (Diagnostic Interview and Structured Hamilton assessment tool), will be used to determine the focus of the emotional response portion of the intervention.

iii. Self-Management Behaviors (SMB) Finally, the Care Coach will discuss patient's self-management behaviors for their comorbidities. He/she will ask the patient to explain how he/she manages each condition, and any challenges he/she faces in self-management.

For example: "Can you describe to me how you manage your COPD? How about your hypertension?" The Care Coach will use the participant's responses, combined with self-reported and objective medication adherence from the observational study, to determine the focus of the SMB portion of 2nd session.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the pilot study if they meet any of the following criteria:

* Low medication adherence for COPD, hypertension, or diabetes medications (score <4.5 on the Medication Adherence Rating Scale, or adherence rate <70% as measured by electronic dose monitoring at study month 15);
* Endorsement of any maladaptive illness belief on the Brief Illness Perceptions Questionnaire for COPD, HTN, or DM;
* Endorsement of any maladaptive medication belief on the Brief Medication Questionnaire for COPD, HTN, or DM.

Exclusion Criteria:

* Adequate medication adherence for COPD
* Adequate medication adherence for hypertension
* Adequate medication adherence for diabetes medications

Score ≥4.5 on Medication Adherence Rating Scale, or adherence rate ≥70% as measured by electronic dose monitoring at Study Month 15.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Brief Illness Perception Questionnaire (BIPQ) | 4 Weeks
  A nine-item scale designed to rapidly assess the cognitive and emotional representations of illness. Full scale range 0 to 10. A higher score reflects a more threatening view of the illness.
Beliefs about Medicines Questionnaire (BMQ scores) | 4 Weeks
  The BMQ assess beliefs about medications. The BMQ has two components: beliefs about overuse (score range from 3-15) and perceived risk of medicines (score range from 5-25), total scale 8-40, higher score indicates stronger beliefs in the concepts of the scale.

SECONDARY OUTCOMES:
Medication Adherence Rating Scale (MARS) | 4 Weeks
  Medication Adherence Rating Scale (MARS) to assess asthma, diabetes, hypertension beliefs about asthma, diabetes and hypertension medication adherence. MARS is a 10-item self-reported instrument. Total scores range from 0 (low likelihood of medication adherence) to 10 (high likelihood), with higher score indicating higher likelihood of medication adherence.
Dietary Approaches to Stop Hypertension (DASH-Q) | 4 Weeks
  The Dietary Approaches to Stop Hypertension (DASH-Q) score examines a dietary pattern and examines relations with health outcomes. The overall score ranges from 8 (the lowest adherence) to 40 (the highest adherence).
International Physical Activity Questionnaire (IPAQ) | 4 Weeks
  The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity. The IPAQ results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Illness Perceptions Questionnaire (IPQ scores) | 4 Weeks
  Multi-factorial pencil-and-paper questionnaire which assesses the five cognitive illness representations on a five-point Likert scale. A revised version of this scale, the Illness Perception Questionnaire- Revised (IPQ-R), extended the original scale by adding more items, splitting the control dimension into personal control and treatment control, and incorporating a cyclical timeline dimension, an overall comprehension of illness factor, and an emotional representation. The IPQ is an 80-item instrument, total scale from 0-10, with higher score indicating higher perception of effects on illness.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Wisnivesky, MD, DrPH, Principal Investigator — Icahn School of Medicine at Mount Sinai; Alex Federman, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No